CLINICAL TRIAL: NCT03402347
Title: Ex Vivo Evaluation of Laser Induced Thermal Tissue Damage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RSP Systems A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RSP-11
Record Dates: First submitted 2018-01-10; First posted 2018-01-18 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-07

CONDITIONS: Gastric Bypass Surgery
Keywords: Ex vivo; Gastric bypass
MeSH Terms: interventions — Radiation, Nonionizing

STUDY DESIGN:
Intervention Model Description: Excess skin from corrective surgery will be evaluated ex vivo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Laser irradiation regimes (Experimental): Non-ionising radiation intervention will be applied to skin explants
  Interventions: Radiation: Non-ionising radiation

INTERVENTIONS:
Radiation: Non-ionising radiation — Laser regimes will be applied to ex vivo skin samples.

SUMMARY:
This clinical study has been initiated to assess the effect of laser exposure on human skin and determine the threshold for tissue damage. The tissue specific effects will be evaluated through histological evaluation. Excess skin from corrective surgery (gastric bypass or similar) will be donated for this study. Skin samples will be subjected to titrating laser treatment with varying laser intensity and exposure time.

DETAILED DESCRIPTION:
The dosimetry of laser induced hyperthermia and threshold for tissue damage will be evaluated. A dose escalation study will be performed by varying irradiance (mW) and time (minutes). Surface temperature will be monitored concurrently. Acute lesions occurring within 5 minutes of irradiation will be assessed and histological damage will be observed microscopically in slice sections of punch biopsies and qualitative assessed. Irradiation regimes above the anticipated threshold will be employed to properly titrate the irradiation necessary to elicit a thermal damage response.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subject 18 years of age or older
* Gastric bypass operated or similar
* Excess abdominal skin to be removed surgically
* Abdominal skin tone 4 or below

Exclusion Criteria:

* Extensive skin changes, tattoos or diseases on skin explant to be donated
* Medical history or any condition that may in investigator's opinion compromise the subject's ability to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-06-16 (Actual); Study Completion 2019-06-16 (Actual)

PRIMARY OUTCOMES:
Thermal damage threshold | Within 3 months
  Quantitative evaluation of laser induced damage by histological lesion in epidermis and dermis.

CONTACTS AND LOCATIONS:
Overall Officials: Jens Ahm Sørensen, MD, Principal Investigator — Department of plastic surgery Z OUH
Locations (1):
- Department of plastic surgery Z OUH, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No